CLINICAL TRIAL: NCT01053052
Title: A Comparative Study of Methods for Tubal Patency Determination and Uterine Cavity Evaluation: Sonography With the FemVue(TM) Catheter System vs. Hysterosalpingography (HSG)
Brief Title: Study of FemVue(TM) Sono Tubal Evaluation System Method Comparison to HSG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled without recruitment
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Femasys 300-001
Record Dates: First submitted 2010-01-18; First posted 2010-01-21 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Fallopian Tube Patency Tests
Keywords: Patency Tests, Fallopian Tubes; Hysterosalpingography; Sonography, Medical
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sonography with FemVue vs. HSG (Experimental): FemVue sonography and HSG
  Interventions: Device: Sonography with FemVue, and HSG

INTERVENTIONS:
Device: Sonography with FemVue, and HSG — Sono HSG for FDA 510(k) cleared indication for use

SUMMARY:
Multi-center prospective comparison of fallopian tubal patency determination and uterine evaluation interventions using legally marketed devices for their intended purposes, and using each subject as their own control.

DETAILED DESCRIPTION:
Study cancelled prior to recruitment.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant women between the ages of 18 and 45 who desire to know the patency status of the fallopian tubes and if the uterine cavity is free of pathology who have:

* Been attempting conception for 6 months or
* A history of PID (including the conditions listed below) or

  * Chlamydia
  * Gonorrhea
  * Endometriosis
* A history of pelvic surgery or
* Advanced maternal age (≥ 35) And
* Negative test for Gonorrhea/Chlamydia or prophylactic antibiotic treatment
* Without current bi-lateral tubal sterilization
* Signed Informed Consent

Exclusion Criteria:

Uterine anomaly or lesion(s) preventing catheter placement for either the FemVue or HSG procedure(as identified and documented by TVUS Screening procedure or the uterine cavity evaluation during the FemVue procedure or any previous diagnostic procedure)

* obstructing access to uterine cornu
* distorting fundus at the midline region

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Concordance of evaluations of fallopian tube patency and intrauterine pathology. | Day 1

SECONDARY OUTCOMES:
subject discomfort assessment | Day 1

IPD SHARING:
Plan to Share IPD: No